CLINICAL TRIAL: NCT01279577
Title: Double-blind, Randomised, Placebo-controlled, Multi-centre Phase II Study to Evaluate the Efficacy and Safety of Three Different Dosages of Oral Trichuris Suis Ova (TSO) Suspension in Active Crohn's Disease
Brief Title: Trichuris Suis Ova (TSO) Suspension Versus Placebo in Active Crohn's Disease
Acronym: TRUST-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSU-2/CDA; 2006-000720-13 (EudraCT Number)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Crohn´s Disease
Keywords: Crohn´s disease; Trichuris suis; randomized; placebo; induction of remission; porcine whipworm
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose TSO (Experimental): Low dose suspension of TSO
  Interventions: Drug: Low dose TSO
- Medium dose TSO (Experimental): Medium dose suspension of TSO
  Interventions: Drug: Medium dose TSO
- High dose TSO (Experimental): High dose suspension of TSO
  Interventions: Drug: High dose TSO
- Placebo (Placebo Comparator): Placebo solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose TSO — Low dose TSO suspension
  Arms: Low dose TSO
Drug: Medium dose TSO — Medium dose TSO suspension
  Arms: Medium dose TSO
Drug: High dose TSO — High dose TSO suspension
  Arms: High dose TSO
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
This study will run in centers in Germany, Denmark, Austria, Czech Republic, and Switzerland, only.

This proof-of-concept study aims to evaluate the efficacy of three doses of oral TSO suspension vs. placebo for the induction of remission in Crohn's disease.

ELIGIBILITY:
Major Inclusion Criteria:

* Signed informed consent,
* Man or woman between 18 and 75 years of age,
* Established diagnosis of Crohn's disease (CD) since at least 3 months prior to screening confirmed by endoscopic and histological, or endoscopic and radiological criteria,
* Negative pregnancy test in females of childbearing potential.

Major Exclusion Criteria:

* Bowel surgery within the last 3 months prior to baseline,
* Resection of more than 50 cm of the ileum,
* Ileostomy or colostomy,
* Septic complications,
* Evidence of infectious diarrhoea (i.e., pathogenic bacteria or Clostridium difficile toxin in stool culture),
* Abscess, perforation, fistulas, or perianal lesions,
* Immediate surgery required (e.g., major stenosis, serious bleeding, peritonitis, ileus),
* Clinical signs of stricturing disease,
* Parenteral or tube feeding,
* Abnormal hepatic function (ALT or ALP > 2.5 x upper limit of normal [ULN] at screening), liver cirrhosis, or portal hypertension,
* Abnormal renal function (Cystatin C > ULN) at screening,
* Any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder, which in the opinion of the investigator might have an influence on the patient's compliance or the interpretation of the results,
* Any condition associated with significant immunosuppression,
* Active malignancy or treatment with anticancer drugs during the last 5 years.
* Existing or intended pregnancy or breast-feeding,
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2010-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rate of clinical remission at week 12 (LOCF) defined as a CDAI< 150 | 12 weeks

SECONDARY OUTCOMES:
Reduction of > 100 points in CDAI | 12 weeks
Adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Schölmerich, Prof., Principal Investigator — Klinikum der Johann Wolfgang Goethe-Universität
Locations (1):
- Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt a.M., Hesse, Germany